CLINICAL TRIAL: NCT04744051
Title: ATCell™ Expanded Autologous, Adipose-Derived Mesenchymal Stem Cells Deployed Via Intravenous Infusion for the Treatment of Post Concussion Syndrome (PCS) in Retired Military and Athletes
Brief Title: ATCell™ Expanded Autologous, Adipose-Derived Mesenchymal Stem Cells Deployed Via Intravenous Infusion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American CryoStem Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRYO_PCS_ADSC_001; FDA File No. 019089 (Other: US Food and Drug Administration)
Record Dates: First submitted 2020-12-15; First posted 2021-02-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Post-Concussion Syndrome
Keywords: Concussion; Adipose Derived Stem Cell; Mesenchymal Stem Cell; Adult Stem Cell; Traumatic Brain Injury; Athletes; Military; Chronic Concussion Syndrome; Post Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The proposed study is a single-site, double-blinded, placebo-controlled study involving a single administration of either individual, autologous ATCell™ lines suspended in 5% dextrose lactated Ringer's solution or a vehicle (5% dextrose lactated Ringer's solution) not containing cells. Each ATCell™ cell line will be created from cells grown from the stromal vascular fraction (SVF) of a participant's own adipose tissue collected by liposuction, and each treated participant will only receive their own cells.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Upon receipt of the harvested tissue sample at the processing facility, eligible participants will be randomized in a one in four ratio to either the 50 million, 150 million or 300 million Adipose derives mesenchymal stem cell (ADMSC) dosage or Placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50 million cell infusion (Active Comparator): Each participant in this arm will receive a single dose of 50 million cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour.
  Interventions: Drug: 50 Adipose Derived Stem Cell Infusion
- 150 million cell infusion (Active Comparator): Each participant in this arm will receive a single dose of 150 million cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour.
  Interventions: Drug: 150 Adipose Derived Stem Cell Infusion
- 300 million cell infusion (Active Comparator): Each participant in this arm will receive a single dose of 300 million cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour.
  Interventions: Drug: 300 Adipose Derived Stem Cell Infusion
- Placebo (Placebo Comparator): Each participant in this arm will receive a single dose of placebo. Upon completion of the study each placebo participant with be given the option to be treated with their cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour. Dosage for the crossover will be determined by the PI following review of data collected from the other arms of the study.
  Interventions: Drug: Placebo Infusion

INTERVENTIONS:
Drug: 50 Adipose Derived Stem Cell Infusion — Each participant in this arm will receive a single dose of 50 million cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour.
  Other Names: Autologous Adipose Derived Mesenchymal Stem Cells; ADSC Infusion Therapy 50
  Arms: 50 million cell infusion
Drug: 150 Adipose Derived Stem Cell Infusion — Each participant in this arm will receive a single dose of 150 million cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour.
  Other Names: Autologous Adipose Derived Mesenchymal Stem Cells; ADSC Infusion Therapy 150
  Arms: 150 million cell infusion
Drug: 300 Adipose Derived Stem Cell Infusion — Each participant in this arm will receive a single dose of 300 million cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour.
  Other Names: Autologous Adipose Derived Mesenchymal Stem Cells; ADSC Infusion Therapy 300
  Arms: 300 million cell infusion
Drug: Placebo Infusion — Each participant in this arm will receive a single dose of placebo. Upon completion of the study each placebo participant will with be given the option to be treated with their cultured adipose derived stem cells derived from their own adipose (fat) tissue via infusion therapy delivery over the course of one hour. Dosage for the crossover will be determined by the PI following review of data collected from the other arms of the study.
  Other Names: ADSC Infusion Therapy Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 Clinical Safety Study intended to provide preliminary assessments of the safety, tolerability, and clinical alleviation of symptoms associated with Post Concussion Syndrome (PCS), also known as Chronic Concussive Syndrome (CCS).

DETAILED DESCRIPTION:
The proposed study is a single-site, double-blinded, placebo-controlled study involving a single administration of either individual, autologous ATCell™ lines suspended in 5% dextrose lactated Ringer's solution or a vehicle (5% dextrose Lactated Ringer's solution) not containing cells. Each ATCell™ cell line will be created from cells grown from the stromal vascular fraction (SVF) of a participant's own adipose tissue collected by liposuction, and each treated participant will only receive their own cells.

Within the treated group, 3 dosing levels will be explored: 50 million cells, 150 million cells, or 300 million cells, and a Placebo group which will receive 5% dextrose lactated Ringer's solution free of cells. Participant follow-ups will take place 1 day following the tissue harvest procedure and, 1 day, 1 week, 1 month, 3 months, and 6 months following ATCell™ treatment. Comprehensive participant's evaluations involving data collection will take place 1, 3, and 6 months following treatment.

It has been proposed that in general, mild traumatic brain injuries (TBI) events need to be taken far more seriously, and that even mild TBI events can result in lasting negative consequences as evidenced by lower performances on neuropsychological assessments when compared with age-matched controls2. In fact, this condition may eventually lead to Alzheimer's Disease (AD) as well as Chronic Traumatic Encephalopathy (CTE), which, together may be termed the AD-like dementias3, further underscoring the need for effective clinical intervention. Currently, no effective treatments are available for this condition aside from treatment of the symptoms, although some more comprehensive treatments have been proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Reviewed and personally signed and dated informed consent document indicating that the participant (or legally acceptable representative) has been informed of and understands all pertinent aspects of the study.
2. Confirmed Diagnosis of Chronic Concussive Syndrome/Post-Concussive Syndrome: At least three (3) of the following criteria must be met to confirm diagnosis:

   A. Persistent headaches

   B. Persistent dizziness

   C. Persistent fatigue

   D. Irritability, intolerance to stress, or unusual emotional reactions

   E. Lowered tolerance to noise and/or light

   F. Impaired memory or concentration

   G. Insomnia
3. Female participants of child bearing potential and at risk of pregnancy during the study must agree to use 2 highly effective methods of contraception throughout the study and for 112 days after the last study visit.
4. Female participant who are not of childbearing potential (i.e. must meet at least one (1) of the following criteria):

   i) Have undergone a documented hysterectomy and/or bilateral oophorectomy

   ii) Have medically confirmed ovarian failure

   iii) Achieved postmenopausal status defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or psychological cause and have a serum follicle stimulating hormone (FSH) level confirming the post menopausal state
5. Individuals who are willing and able to comply with lifestyle guidelines, scheduled visits, treatment plan, laboratory tests, and other study procedures through the end of the final study visit
6. Individuals Aged 18 to 65 at the time of screening and enrollment.

Exclusion Criteria:

1. Any cardiac pathologies or conditions which may risk the participant or interfere with the ability to interpret the results. Signs and symptoms of clinically significant cardiac disease including but not limited to:

   A. Ischemic cardiac disease (eq. unstable angina, myocardial infarction) in the 6 months prior to screening.

   B. New York Heart Association (NYHA) Class III or IV congestive heart failure or known left ventricular dysfunction with ejection fraction ≤ 35%, cardiomyopathy, myocarditis in the 6 months prior to screening.

   C. Resting tachycardia (heart rate ≥ 120) or resting bradycardia (heart ≤ 45) on ECG at screening.

   D. Any other cardiovascular illness that in the opinion of the Investigator would render an individual unable to participate in the study.

   E. Individuals with history of heart block.

   F. Individuals with a history of Atrial Fibrillation

   G. Individuals that have had stents implanted within one year of recruitment
2. History of transient ischemic attack in the 6 months prior to screening, diagnosis of stroke with residual deficits (eq. aphasia, substantial motor or sensory deficits) diagnosis of stroke with residual deficits (eq. aphasia, substantial motor or sensory deficits) that would preclude completion of required study activities
3. Resting, sitting blood pressure (BP) ≥ 160 mm Hg in systolic pressure or ≥ 100 mm Hg in diastolic pressure at screening. If a participant is found to have untreated significant hypertension at screening and antihypertensive treatment is initiated, assessment for study eligibility should be deferred until BP and antihypertensive medication have been stable for at least 1 month. For participants with previously diagnosed hypertension, antihypertensive medications must be stable for at least 1 month prior to screening
4. Participants who have evidence of orthostatic hypotension based upon replicate orthostatic blood pressure measurements. If orthostatic blood pressure change is not able to be determined (e.g., unable to establish a stable supine systolic and diastolic blood pressure) the participant is not eligible for the study
5. Individuals with a history of Deep Vein Thrombosis (DVT) or pulmonary embolism
6. Individuals with a history or family history of thrombophilia such as Factor V Leiden
7. Individuals that have had stents implanted within the past year
8. Individuals that are currently being treated with an anticoagulant medication
9. History, diagnosis, or signs and symptoms of clinically significant neurological disease, including but not limited to:

   A. Alzheimer's disease or other type of dementia

   B. Peripheral or autonomic neuropathy

   C. Multiple sclerosis

   D. Epilepsy or seizure disorder with history of seizure within the last 2 years

   E. Myopathy

   F. White matter disease
10. Individuals currently being treated with specific prescription immunomodulatory agents:

    A. Certolizumab (Cimzia™)

    B. Infliximab (REMICADE™)

    C. Etanercept (Enbrel™)

    D. Prednisone (Deltasone, Rayos, Prednisone Intensol)

    E. Prednisolone (Omnipred™)

    F. Dexamethasone (Ozurdex™)

    G. Any drug which the investigator believes would compromise the results or interfere with ATCell™ effectiveness
11. Participant with any active or chronic infection
12. Life-threading organ dysfunction
13. Planned surgical procedure during the duration of the study
14. Largely or wholly incapacitated (eq. individual bedridden or confined to wheelchair, permitting little or no self care)
15. Pregnant or actively breastfeeding females; females of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study, meaning 6 months after ATCell™ administration
16. Severe physical limitations or disabilities
17. Participants who are seropositive for Human Immunodeficiency Virus -1 (HIV1), Human Immunodeficiency Virus -2 (HIV2), Hepatitis B Surface Antigen and Hepatitis C, indicative of current infection
18. Participant unable to give written consent in accordance with institutional review board guidelines
19. Treatment with any immunosuppressive therapy within 3 months of evaluation
20. Current or recent treatment (within 3 months of evaluation) with an investigational drug and/or therapy (phase 1-4) within 90 days of screening
21. Individuals with a concurrent diagnosis of malignant neoplasm (cancer)
22. History of cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
23. Individuals with inadequate subcutaneous tissue to allow for appropriate lipoaspirate collection
24. Other severe or chronic medical psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make this individual inappropriate for entry into this study
25. Individuals with immunodeficiencies or severe autoimmune disease
26. Individuals allergic to local anesthetics
27. Individuals with any contraindication to liposuction, in the investigator's opinion
28. History of coagulation disorders that would put them at risk
29. Individuals, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason
30. The individual is involved in an active civil, criminal or workers compensation case other than the NFL class action
31. Individuals unable or unwilling to return for the required follow-up evaluations
32. Presence of drugs of abuse (including cannabis and prescription medications without valid prescription), or illegal drugs in the urine toxicology test obtained at screening
33. History of known alcohol, analgesic or drug abuse within 2 years of screening
34. Individuals who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or who are employees directly involved in the conduct of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Health Status using the 36 item Short Form Health Survey (SF-36) | Baseline, 1 month and 6 months post treatment
  Completed by Participant as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores of completed SF-36 will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative).The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Assessment of Visual Attention and Task Switching | Baseline, 1 month and 6 months post treatment
  Administered by study staff as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores How long it takes the participant to connect a sequence of 25 consecutive targets in sequential order on a sheet of paper or computer screen to complete the two tests will be numerically determined (seconds) and compared to baseline. The goal of the test is for the subject to finish both parts as quickly as possible, with the time taken to complete the test being used as the primary performance metric If a person makes an error in the test, there's no change in the score other than that it makes their completion time longer since the person has to go back to correct the error, thus extending their time, shorter completion times indicate improved scores.
Assessment of Contextual Verbal Learning | Baseline, 1 month post treatment and 6 months post treatment
  Administered by study staff as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative)
Assessment of Verbal Fluency | Baseline, 1 month post treatment and 6 months post treatment
  Administered by study staff as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative). Scoring is based on total word numbers (expressed in 60 seconds), higher totals in tests indicate improvement
Assessment of Attention and Executive functions | Baseline, 1 month post treatment and 6 months post treatment
  Administered by study staff as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined as the number of correct answers provided in 90 seconds. and compared to baseline. Changes against baseline will be represented numerically (positive or negative). AN increase in total correct answers will indicate improvement
Assessment of Unstructured Verbal Learning and Memory | Baseline, 1 month post treatment and 6 months post treatment
  Administered by study staff as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined based the total number of correct answers in 3 categories of 12 and compared to baseline as a percentage. Changes against baseline will be represented numerically (positive or negative), Improved scores will indicate improvement.
Assessment of Visuospatial Learning and Memory | Baseline, 1 month post treatment and 6 months post treatment
  Administered by study staff as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined (percent) based upon correct recall and compared to baseline. Changes against baseline will be represented numerically (positive or negative).
Assessment of Symptoms of Anxiety over Time | Baseline, 1 month post treatment and 6 months post treatment
  Completed by Participant as a part of physician visits at baseline, and 1, and 6 months following treatment. Each question is scored on a scale of 1 to 4 for 22 questions, total score is the sum of the score of each item (1-4) will be numerically determined and compared to baseline. Changes against baseline will be represented numerically (positive or negative). Lower scores will indicate improvement.
Assessment of Pain | Baseline, 1 month post treatment and 6 months post treatment
  Completed by Participant as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined on a scale of 1 to 10 and compared to baseline. Changes against baseline will be represented numerically (positive or negative) lower scores will indicate improvement.
Assessment of Sleep Quality | Baseline, 1 month post treatment and 6 months post treatment
  Completed by Participant as a part of physician visits at baseline, and 1, and 6 months following treatment. Scores will be numerically determined (1 to 3) for 7 questions (maximum score of 21) and compared to baseline. Changes against baseline will be represented numerically (positive or negative). Lower total scores indicate improvement.
Assessment of Treatment by Participant | Baseline, 1 month post treatment and 6 months post treatment
  Completed by Participant as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined on a 1 to 7 basis, and compared to baseline. Changes against baseline will be represented numerically (positive or negative) lower scores represent improvement.
Assessment of Depression by Participant | Baseline, 1 month post treatment and 6 months post treatment
  Completed by Participant as a part of physician visits at baseline, and 1, and 6 months following treatment . Scores will be numerically determined (1 to3) for 9 questions (maximum score of 27) and compared to baseline. Changes against baseline will be represented numerically (positive or negative), lower scores indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Hanson, MD, Principal Investigator — Biosolutions Clinical Research Center
Locations (1):
- BioSolutions Clinical Research Center, La Mesa, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein MB, Ursano RJ, Campbell-Sills L, Colpe LJ, Fullerton CS, Heeringa SG, Nock MK, Sampson NA, Schoenbaum M, Sun X, Jain S, Kessler RC. Prognostic Indicators of Persistent Post-Concussive Symptoms after Deployment-Related Mild Traumatic Brain Injury: A Prospective Longitudinal Study in U.S. Army Soldiers. J Neurotrauma. 2016 Dec 1;33(23):2125-2132. doi: 10.1089/neu.2015.4320. Epub 2016 Apr 8. PMID 26905672
- [Background] Sterr A, Herron KA, Hayward C, Montaldi D. Are mild head injuries as mild as we think? Neurobehavioral concomitants of chronic post-concussion syndrome. BMC Neurol. 2006 Feb 6;6:7. doi: 10.1186/1471-2377-6-7. PMID 16460567
- [Background] Ramos-Cejudo J, Wisniewski T, Marmar C, Zetterberg H, Blennow K, de Leon MJ, Fossati S. Traumatic Brain Injury and Alzheimer's Disease: The Cerebrovascular Link. EBioMedicine. 2018 Feb;28:21-30. doi: 10.1016/j.ebiom.2018.01.021. Epub 2018 Jan 31. PMID 29396300
- [Background] McKee AC, Robinson ME. Military-related traumatic brain injury and neurodegeneration. Alzheimers Dement. 2014 Jun;10(3 Suppl):S242-53. doi: 10.1016/j.jalz.2014.04.003. PMID 24924675
- [Background] Thompson M, Mei SHJ, Wolfe D, Champagne J, Fergusson D, Stewart DJ, Sullivan KJ, Doxtator E, Lalu M, English SW, Granton J, Hutton B, Marshall J, Maybee A, Walley KR, Santos CD, Winston B, McIntyre L. Cell therapy with intravascular administration of mesenchymal stromal cells continues to appear safe: An updated systematic review and meta-analysis. EClinicalMedicine. 2020 Jan 17;19:100249. doi: 10.1016/j.eclinm.2019.100249. eCollection 2020 Feb. PMID 31989101
- [Background] Toyserkani NM, Jorgensen MG, Tabatabaeifar S, Jensen CH, Sheikh SP, Sorensen JA. Concise Review: A Safety Assessment of Adipose-Derived Cell Therapy in Clinical Trials: A Systematic Review of Reported Adverse Events. Stem Cells Transl Med. 2017 Sep;6(9):1786-1794. doi: 10.1002/sctm.17-0031. Epub 2017 Jul 19. PMID 28722289